CLINICAL TRIAL: NCT01078428
Title: Effect of Transparent, Self-drying Silicone Gel on the Treatment of Hypertrophic Abdominal Scars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Woraphong Manuskiatti, M.D., Professor, Mahidol University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Si 193/2009; 125/2552(EC4) (Other: Siriraj Institutional Review Board)
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Keloids; Hypertrophic Scars
Keywords: Hypertrophic scars; Topical silicone gel; Scar thickness; Scar Color; Scar pliability; Scar appearance
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic | interventions — Silicone Gels; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silicone gel (Active Comparator): Gel containing silicone gel
  Interventions: Other: Topical silicone gel
- Vaseline (Placebo Comparator): Gel containing petrolatum gel
  Interventions: Other: Vaseline

INTERVENTIONS:
Other: Topical silicone gel — Topical silicone gel will be applied to the scar twice daily for a period of 8 weeks
  Other Names: Dermatix gel
  Arms: Silicone gel
Other: Vaseline — Topical petrolatum gel will be applied to the scar twice daily for a period of 8 weeks
  Arms: Vaseline

SUMMARY:
Keloids and hypertrophic scars are a common subject of dermatologic consultations. Therapeutic management of such conditions remains challenging because of their high rate of recurrence and lack of curative treatment.

DETAILED DESCRIPTION:
Silicone gel Sheeting (SGS) is one treatment modality that has proven effective for treatment of hypertrophic scar. One disadvantage of SGS is its application technique. To be effective, SGS must be applied on the scar for at least 12 hours daily. Topical silicone gel is a novel therapy that has shown promising result on scar prevention. However, the efficacy and safety of topical silicone gel for treatment of hypertrophic scar has not been confirmed.

ELIGIBILITY:
Inclusion Criteria:

* subjects at least 18 years old
* subjects with hypertrophic abdominal scar
* Have not received treatment on the scar at least 1 month prior to the enrollment.

Exclusion Criteria:

* subject who has previous history of silicone allergy
* subject who smoke cigarette
* subject who was treated with x-rays irradiation in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Scar thickness | 1, 2 and 5 months after initiation of treatment

SECONDARY OUTCOMES:
Clinical assessment on overall scar appearance | 1, 2 and 5 months after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong - Manuskiatti, M.D., Principal Investigator — Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Kloeters O, Tandara A, Mustoe TA. Hypertrophic scar model in the rabbit ear: a reproducible model for studying scar tissue behavior with new observations on silicone gel sheeting for scar reduction. Wound Repair Regen. 2007 Sep-Oct;15 Suppl 1:S40-5. doi: 10.1111/j.1524-475X.2007.00224.x. PMID 17727466
- [Background] Murison M, James W. Preliminary evaluation of the efficacy of dermatix silicone gel in the reduction of scar elevation and pigmentation. J Plast Reconstr Aesthet Surg. 2006;59(4):437-9. doi: 10.1016/j.bjps.2005.09.037. No abstract available. PMID 16756266
- [Background] Chan KY, Lau CL, Adeeb SM, Somasundaram S, Nasir-Zahari M. A randomized, placebo-controlled, double-blind, prospective clinical trial of silicone gel in prevention of hypertrophic scar development in median sternotomy wound. Plast Reconstr Surg. 2005 Sep 15;116(4):1013-20; discussion 1021-2. doi: 10.1097/01.prs.0000178397.05852.ce. PMID 16163087
- [Background] Li-Tsang CW, Lau JC, Choi J, Chan CC, Jianan L. A prospective randomized clinical trial to investigate the effect of silicone gel sheeting (Cica-Care) on post-traumatic hypertrophic scar among the Chinese population. Burns. 2006 Sep;32(6):678-83. doi: 10.1016/j.burns.2006.01.016. Epub 2006 Jul 11. PMID 16837136